CLINICAL TRIAL: NCT01883947
Title: Touch Massage in the Sub-acute Phase After Stroke - Does it Have Impact on General Health and Independence?
Brief Title: Effects of Touch Massage in the Sub-acute Phase After Stroke
Acronym: MEST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: too long inclusion phase due to difficulties to find eligible participants.
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Kristina Lämås, PhD, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2012-494-32M
Record Dates: First submitted 2013-05-27; First posted 2013-06-21 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Stroke
Keywords: Stroke; Massage; General Health; Independence
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Touch massage (Experimental): Intervention group will receive touch massage on hands and feet and the intervention will start one week after the onset of stroke and last for 30 minutes each time, five days a week for two weeks
  Interventions: Procedure: Touch massage
- non-TENS (Sham Comparator): The sham treatment will start one week after the onset of stroke and last for 30 minutes each time, five days a week for two weeks
  Interventions: Other: non-TENS

INTERVENTIONS:
Procedure: Touch massage — Touch massage is a gentle massage with strokes on hands, arms, feet and legs with at pressure of 2.5 N which is more gentle than Swedish massage but harder than strokes performed with a brush. The speed of the strokes is about 1-5 cm/sec. During the massage, the subjects will lie on a bed. Intervention group will receive touch massage on hands and feet and the intervention will start one week after the onset of stroke and last for 30 minutes each time, five days a week for two weeks
  Arms: Touch massage
Other: non-TENS — Subjects in the control group will have sham treatment which is a non-active transcutaneous electrical nerve stimulation (non-TENS), while they lie in bed with electrodes attached to the skin of the affected arm. The device will be manipulated in a way so that no electrical impulses will reach the electrodes. During treatment, the masseur will remain in the room without initiating any conversation.
  Arms: non-TENS

SUMMARY:
The aim is to study effects of touch massage in the sub-acute phase after stroke in two main areas; general health and independence.The hypothesis are that; touch massage in the sub-acute phase after stroke decreases anxiety and pain, increases health related-quality of life, decrease physiological stress responses, increase sensorimotor function, decrease disability, and increase activity in sensorimotor areas and decrease redundant brain activity in motor-related areas.

DETAILED DESCRIPTION:
Despite high quality stroke care in Sweden, decreased sensorimotor function, anxiety and pain remains one year after stroke and lead to impaired health and dependence as well as high health care costs. It is therefore urgent to find new rehabilitation strategies. There is some knowledge about effects of touch massage among healthy and patients with ill-health conditions but no study have evaluated touch massage in the sub-acute phase of stroke. Therefore the aim in this project is to study effects of t touch massage in the sub-acute phase after stroke in two main areas; general health and independence.

ELIGIBILITY:
Inclusion Criteria:

* stroke defined according to Trial of ORG 10172 in Acute Stroke Treatment (TOAST) and The Oxford Community Stroke Project Classification (OSPC),
* impaired finger tapping on the affected side of the body,
* the ability to flex the wrist 20° from substrate on affected side of the body

Exclusion Criteria:individuals with

* cancerous tumors,
* infections with fever,
* neurologic or psychiatric disease,
* alcohol or drug addiction,
* conditions that impede communication.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-01; Primary Completion 2017-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Scale | 2 month
  Assessment of self-rated anxiety on two subscales. Traits are stable over time and not sensitive to occasional stressors. States are sensitive for occasional stressors assessing current emotional state

SECONDARY OUTCOMES:
VAS | 2 weeks
  To assess self-rated pain
Nottingham Health Profile | 2 weeks
  This is a self-rating scale which assess Health related quality of life
ECG | 2 weeks
  evaluate heart rate variability which reflects activity in the autonomic nervous system
Salivary cortisol | 2 weeks
  To assess effects on stress responses
Blood pressure | 2 weeks
  to assess effects on stress responses
Shape Texture Identification Test | 2 month
  will be used to assess touch discrimination
Box and Blocks | 2 month
  will be used to test gross dexterity
Nine Hole Peg | 2 month
  will be used to test fine motor dexterity,
Jamar® Hydraulic Hand Dynamometer | 2 month
  will be used to assess grip strength
movement laboratory with high-speed cameras | 2 month
  Temporal and spatial kinematic variables will be evaluated
Functional magnetic resonance imaging | 2 weeks
  Evaluation of brain activity while patient perform finger-tapping/movement with the paretic hand
Barthel index and Modified Ranking scale | 2 month
  will be used to assess disability after stroke

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Lämås, PhD, Principal Investigator — Umea University
Locations (1):
- Norrlands university hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lamas K, Hager C, Lindgren L, Wester P, Brulin C. Does touch massage facilitate recovery after stroke? A study protocol of a randomized controlled trial. BMC Complement Altern Med. 2016 Feb 4;16:50. doi: 10.1186/s12906-016-1029-9. PMID 26846253